CLINICAL TRIAL: NCT04833998
Title: Hydration Based on Thoitaine, Aloe Vera and Calendula, in the Prevention of Hand-Foot Syndrome in Patients Using Capecitabine: TACX Care Trial
Brief Title: Hydration Based on Thoitaine, Aloe Vera and Calendula, in the Prevention of Hand-Foot Syndrome in Patients Using Capecitabine
Acronym: TACX Care
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Brasileiro de Controle do Cancer (Other)
Collaborators: Wecare Comércio de Cosméticos (Unknown)
Responsible Party: Principal Investigator, Flavia Viecili Tarcha, Principal Investigator, Instituto Brasileiro de Controle do Cancer
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 01629018.1.0000.0072
Record Dates: First submitted 2021-03-30; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Hand-foot Syndrome
Keywords: Hand-foot Syndrome; Palmoplantar Erythrodysesthesia; Acral Erythema; Capecitabine; Moisturizing cream
MeSH Terms: conditions — Hand-Foot Syndrome

STUDY DESIGN:
Intervention Model Description: The allocation ratio is 2:1, favouring the active treatment. In this study we are using unequal allocation ratios for a variety of reasons, including allowance for learning curves, and ethical considerations when the balance of existing evidence appears to be in favour of one intervention over the placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo will be cream without the active ingredient. It will be matched in appearance, smell, consistency, and color to Extremecare topical cream. Patients will be instructed to apply the placebo cream to the hand and feet.
  Interventions: Drug: Placebo
- Extremecare (Experimental): Extremecare is a moisturizing cream based on Thoitaine, Aloe Vera and Calendula for topical use. Patients will be instructed to apply the moisturizing cream to the hand and feet.
  Interventions: Drug: Extremecare

INTERVENTIONS:
Drug: Extremecare — The product under investigation (Extremecare) will be supplied as 120g use individual tubes to be applicated in the hands and feet twice a day (once in the morning and once in the evening) beginning with the first cycle of capecitabine and continuing until the end of the fifth cycle of chemotherapy.
  Arms: Extremecare
Drug: Placebo — Placebo cream will be supplied as 120g use individual tubes to be applicated in the hand and feet twice a day (once in the morning and once in the evening) during the fifth cycle of capecitabine therapy.
  Arms: Placebo

SUMMARY:
Hand-foot syndrome (HFS) is a very common adverse event of many chemotherapeutic agents, especially capecitabine. The HFS can considerably interfere patient quality of life (QoL).

The current treatments for hand-foot symptoms no have demonstrated 100% efficacy. And, the dose reduction and treatment interruption are recommended for treatment of HFS.

It is known that hydration improves the degree of hand-foot syndrome, as it improves moisture retention and maintain hydration, thereby reducing further desquamation and decreasing infection risks. But so far there is no evidence of a cream that improves incidence. Besides that, clinical trials evaluating the use of urea-based moisturizer in patients treated with capecitabine have not shown efficacy in preventing hand-foot syndrome.

The purpose of this study is to evaluate the effectiveness of moisturizer based on Thoitaine, Aloe Vera and Calendula compared to placebo in the prevention of SMP of any degree, in patients using Capecitabine.

DETAILED DESCRIPTION:
The research product, proposed in this study, was developed to meet the specific hydration needs of patients undergoing cancer treatment and is produced from nine main ingredients with natural moisturizing actions based on glycerin, hazelnut extract, shea butter, aloe vera, calendula, chamomile and oat extract and 2 antioxidants (vitamin E and Thoitaine), dermatologically tested and approved. The choice of the product was based, mainly, due to its natural components, whose data from previous studies were extrapolated from radiodermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age
* Patients with gastrointestinal tumors or breast cancer who will be treated with capecitabine
* Indication of adjuvant or palliative treatment with capecitabine
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Information of the patient and signature of the informed consent form by the patient or her legal representative.

Exclusion Criteria:

* Previous chemotherapy with capecitabine
* Pre-existing patients with neuropathies
* Patients with known allergic reactions to any of the ingredients of the investigational product
* Patients with dermatological conditions that affect the hands or feet
* Patients with rectal neoplasia and indication for neoadjuvant treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2019-08-02 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients presenting Hand-foot Syndrome (HFS) any grade secondary to capecitabine therapy. | Up to 15 weeks
  Number of Patients who developed Hand-foot Syndrome (HFS) by Toxicity Grade. The incidence and severity of hand-foot syndrome (HFS) developed during chemotherapy will be defined by using the grading system for HFS per the NCI Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03 for all patients assigned who received at least 1 cycle of capecitabine. Investigators assess and fill the grading into the case report form every visit.

SECONDARY OUTCOMES:
Changes in the signs of hand-foot syndrome | Baseline and 1-2-3-4-5 cycles of capecitabine-containing chemotherapy (each cycle is 21 days)
  Digital Photos will be taken of the hands and feet at 21 day intervals until the fifth cycles of capecitabine-containing chemotherapy ended to evaluate Erythema, desquamation, edema, ulceration, vesicopustules.
Incidence of capecitabine dose modifications (dose delay and dose reductions) due to toxicity. | Up to 15 weeks
  Determined by the number of patients who required a toxicity-related, dose reduction of capecitabine during active treatment at each cycle where a dose reduction occurred
Quality of Life as Measured by Dermatology Life Quality Index (DLQI) | Up to 15 weeks
  Dermatology Life Quality Index (DLQI) consists of 10 questions concerning patients' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week. The DLQI item response options are rated by the participant from 0 (not at all/not relevant) to 3 (very much). The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. It is self explanatory and is usually completed in one or two minutes.
Incidence of cessation of capecitabine therapy | Up to 15 weeks
  Cessation of capecitabine thereby because any toxicity

CONTACTS AND LOCATIONS:
Locations (1):
- IBCC Oncologia, São Paulo, Brazil